CLINICAL TRIAL: NCT00064207
Title: Randomized Phase II/III Study Comparing Gemcitabine Followed by Gemcitabine Plus Concomitant Radiation (50.4 Gy) Versus Control After Curative Pancreaticoduodenectomy for Pancreatic Head Cancer
Brief Title: Gemcitabine and Radiation Therapy Compared With Gemcitabine Alone in Treating Patients Who Have Undergone Surgery for Pancreatic Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-40013-22012; EORTC-40013; EORTC-22012; FFCD-0304; EU-20540
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as gemcitabine use different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving these treatments after surgery may kill any tumor cells that remain after surgery. It is not yet known whether giving gemcitabine together with radiation therapy is more effective than gemcitabine alone following surgery in treating pancreatic cancer.

PURPOSE: This randomized phase II/III trial is studying how well giving gemcitabine together with radiation therapy works and compares it to gemcitabine alone in treating patients who have undergone surgery for pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Phase II:

* Determine the feasibility of gemcitabine followed by chemoradiotherapy with gemcitabine vs gemcitabine alone after prior curative resection in patients with pancreatic head adenocarcinoma.
* Compare the tolerability of these regimens, in terms of acute and late toxicity, in these patients.

Phase III:

* Compare the disease-free and overall survival of patients treated with these regimens .
* Compare the quality of life of patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Determine the sites of recurrence in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to ECOG/WHO performance status (0-1 vs 2), participating center, and N stage (N0 vs N1 vs NX). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Within 8 weeks after prior surgical resection, patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 4 weeks for 2 courses.

Patients then receive additional gemcitabine IV over 30 minutes on days 57, 64, 71, 78, 85, and 92. Beginning on day 57, patients also undergo radiotherapy once daily, 5 days a week, for 6 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

* Arm II: Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 4 weeks for 4 courses.

Quality of life (QOL) is assessed in both arms, according to the following schedules:

* Arm I: QOL is assessed at baseline; at 3 weeks after the beginning of chemoradiotherapy; after the completion of chemoradiotherapy; every 3 months for 2 years; and then every 6 months for 1 year.
* Arm II: QOL is assessed at baseline; at 12 weeks; at 16 weeks; every 3 months for 2 years; and then every 6 months for 1 year.

Patients are followed every 3 months for 2 years and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 538 patients (269 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed pancreatic head adenocarcinoma
* Prior pancreaticoduodenectomy required

  * Documented histological examination of surgical margins (R0), including retroperitoneal margin
  * Performed within the past 8 weeks
* Any number of lymph nodes (less than 10 OR 10 or more) allowed
* No periampullary cancer

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC greater than 3,500/mm^3
* Platelet count greater than 150,000/mm^3
* Hemoglobin greater than 9.0 g/dL

Hepatic

* Bilirubin less than 1.5 times normal
* AST and ALT less than 3.0 times normal

Renal

* Creatinine less than 1.2 mg/dL

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other prior or concurrent malignancy except basal cell skin cancer or carcinoma in situ of the cervix
* No psychological, familial, sociological, or geographical condition that would preclude study compliance and follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy

Chemotherapy

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy

Surgery

* See Disease Characteristics
* Recovered from prior surgery

Other

* No other concurrent anticancer agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2003-05; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of full completion of treatment as measured by the number of patients completing treatment 1 month after treatment in phase II
Tolerability in terms of acute toxicity as measured by NCI-CTC v2.0 1 month after completion of treatment in phase II
Tolerability in terms of late toxicity as measured by EORTC and RTOG 1 month after completion of treatment in phase II
Overall survival as measured by Logrank every 3 months in years 1-2, and every 6 months thereafter in phase III

SECONDARY OUTCOMES:
Disease-free survival as measured by Logrank every 3 months in years 1-2, and every 6 months thereafter
Acute toxicity as measured by NCI-CTC v2.0 every 3 months in years 1-2, and every 6 months thereafter
Late toxicity as measured by EORTC and RTOG every 3 months in years1-2, and every 6 months thereafter
Quality of life as measured by Quality of Life Questionnaire Core 30 (QLQ-C30) v3.0 and EORTC QLQ PAN-26 every 3 months in years 1-2 and every 6 months thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Van Laethem, MD, PhD, Study Chair — Erasme University Hospital; Volker G. Budach, MD, PhD, Study Chair — Charite University, Berlin, Germany; Pascal Hammel, MD, PhD, Study Chair — Hopital Beaujon
Locations (59):
- Belgium (6):
  - Hopital Universitaire Erasme, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Hopital de Jolimont, Haine-Saint-Paul
  - Cazk Groeninghe - Campus St-Niklaas, Kortrijk
  - CHU Liege - Domaine Universitaire du Sart Tilman, Liège
  - Algemeen Ziekenhuis Sint-Augustinus, Wilrijk
- France (45):
  - Centre Hospitalier d'Abbeville, Abbeville
  - Centre Hospitalier d'Annecy, Annecy
  - Institut Sainte Catherine, Avignon
  - Hopital Duffaut, Avignon
  - C.H.G. Beauvais, Beauvais
  - Centre Hospitalier de Blois, Blois
  - Clinique Tivoli, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Boucher
  - Centre Hospitalier Universitaire Ambroise Pare - Boulogne, Boulogne-Billancourt
  - Centre Hospitalier Docteur Duchenne, Boulogne-sur-Mer
  - Centre Hospitalier Pierre Oudot, Bourgoin
  - CHU de Caen, Caen
  - CHR Clermont Ferrand, Hotel dieu, Clermont-Ferrand
  - Hopital Beaujon, Clichy
  - Louis Mourier Hospital, Colombes
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Centre Hospitalier de Dax, Dax
  - Hopital Du Bocage, Dijon
  - Centre Hospitalier Intercommunal St. Aubin les Elbeuf, Elbeuf
  - CHU de Grenoble - Hopital de la Tronche, Grenoble
  - Centre Hospitalier Departemental, La Roche-sur-Yon
  - Clinique Victor Hugo, Le Mans
  - Hopital Robert Boulin, Libourne
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Clinique Saint Jean, Lyon
  - Centre Leon Berard, Lyon
  - CHU de la Timone, Marseille
  - Centre Hospitalier General de Mont de Marsan, Mont-de-Marsan
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Hospitalier de Mulhouse, Mulhouse
  - C.H.U. de Nimes - Groupe Hospitals-Universitaire Caremeau, Nîmes
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Bichat - Claude Bernard, Paris
  - Hopital Saint Antoine, Paris
  - CHU Pitie-Salpetriere, Paris
  - Hopital Cochin, Paris
  - Hopital Tenon, Paris
  - C.H.G. De Pau, Pau
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Poitiers, Poitiers
  - Hopital Charles Nicolle, Rouen
  - Centre Paul Strauss, Strasbourg
  - Hopital Universitaire Hautepierre, Strasbourg
  - Centre Hospitalier Universitaire Bretonneau de Tours, Tours
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
- Germany (5):
  - Charite - Campus Charite Mitte, Berlin
  - Robert Roessle Comprehensive Cancer Center at University of Berlin - Charite Campus Buch, Berlin
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Johannes Gutenberg University, Mainz
  - Munich Oncologic Practice at Elisenhof, Munich
- Rambam Medical Center, Haifa, Israel
- Academisch Medisch Centrum at University of Amsterdam, Amsterdam, Netherlands
- Hopital Cantonal Universitaire de Geneve, Geneva, Switzerland

REFERENCES:
- [Result] Van Laethem JL, Hammel P, Mornex F, Azria D, Van Tienhoven G, Vergauwe P, Peeters M, Polus M, Praet M, Mauer M, Collette L, Budach V, Lutz M, Van Cutsem E, Haustermans K. Adjuvant gemcitabine alone versus gemcitabine-based chemoradiotherapy after curative resection for pancreatic cancer: a randomized EORTC-40013-22012/FFCD-9203/GERCOR phase II study. J Clin Oncol. 2010 Oct 10;28(29):4450-6. doi: 10.1200/JCO.2010.30.3446. Epub 2010 Sep 13. PMID 20837948
- [Result] Van Laethem J, Van Cutsem E, Hammel P, et al.: Adjuvant chemotherapy alone versus chemoradiation after curative resection for pancreatic cancer : feasibility results of a randomised EORTC/FFCD/GERCOR phase II/III study (40013/22012/0304). [Abstract] J Clin Oncol 26 (Suppl 15): A-4514, 2008.